CLINICAL TRIAL: NCT07000812
Title: Neurophysiological Effects of Cognitive Behavioral Therapy in the Treatment of Obsessive-Compulsive Disorder: An EEG Clinical Study
Brief Title: EEG Evaluation of CBT for Obsessive-Compulsive Disorder
Acronym: CBT-OCD-EEG
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Uskudar University (Other)
Collaborators: Istanbul Nisantasi University (Other); Beykoz University (Other)
Responsible Party: Principal Investigator, Selami Varol Ülker, Dr, Uskudar University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 61351342/020-674
Record Dates: First submitted 2025-04-07; First posted 2025-06-03 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-06

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: Cognitive Behavioral Therapy; EEG; Neurophysiology; ERP (Exposure and Response Prevention); OCD
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to one of two parallel groups: CBT treatment group or waiting list control group.
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessor conducting EEG assessments and psychological evaluations is blinded to group assignment. Participants and therapists cannot be blinded due to the nature of the psychotherapy intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CBT Intervention Group (Experimental): Participants receive 12 weekly individual Cognitive Behavioral Therapy (CBT) sessions, each session lasting approximately 50 minutes. CBT includes Exposure and Response Prevention (ERP), cognitive restructuring, psychoeducation, and relapse prevention strategies.
  Interventions: Behavioral: Cognitive Behavioral Therapy (CBT)
- Waiting List Control (No Intervention): Participants receive no intervention during the 12-week treatment period but are offered CBT treatment after the completion of the study.

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy (CBT) — Participants in the intervention arm receive 12 weekly sessions of individual CBT. Therapy includes exposure and response prevention, cognitive restructuring, psychoeducation, and relapse prevention strategies.
  Arms: CBT Intervention Group

SUMMARY:
This clinical trial investigates how Cognitive Behavioral Therapy (CBT), a psychological treatment that helps people change their thought and behavior patterns, affects brain function in people diagnosed with Obsessive-Compulsive Disorder (OCD). OCD is characterized by repeated, unwanted thoughts (obsessions) and behaviors (compulsions) that significantly interfere with daily life.

Although CBT is known to effectively reduce OCD symptoms, exactly how it changes brain activity remains unclear. This study aims to measure the effects of CBT on brain function using electroencephalography (EEG), a safe, non-invasive way to monitor brain activity.

Participants diagnosed with OCD will be randomly assigned to two groups. One group will receive CBT consisting of 12 individual therapy sessions, held weekly, lasting about 50 minutes each. The other group will not receive therapy during the study but will be offered treatment afterward. Brain activity and psychological well-being will be measured three times: before starting treatment, immediately after completing CBT, and again three months later.

By comparing these two groups, the study hopes to answer whether CBT causes measurable changes in brain activity and how these changes relate to improvements in OCD symptoms. Results from this study could help improve future treatments and understanding of OCD.

DETAILED DESCRIPTION:
Obsessive-Compulsive Disorder (OCD) is a psychiatric condition marked by persistent, distressing obsessions (intrusive thoughts) and compulsions (repetitive behaviors aimed at relieving anxiety). Cognitive Behavioral Therapy (CBT), particularly with Exposure and Response Prevention (ERP), is established as an effective treatment method. However, the exact neurophysiological mechanisms underlying CBT-induced symptom improvement in OCD patients remain unclear.

This randomized controlled clinical trial aims to clarify these mechanisms by examining how CBT impacts brain functioning through neurophysiological assessments using electroencephalography (EEG). EEG is a reliable and non-invasive method for measuring brain electrical activity, particularly valuable for observing real-time brain responses to various cognitive tasks and resting-state conditions.

The trial will recruit 60 adult OCD patients (aged 18-65) diagnosed according to DSM-5 criteria from outpatient psychiatric clinics in Istanbul, Turkey. After baseline assessments, participants will be randomly assigned equally into two groups:

Intervention Group (CBT): Participants will receive 12 weekly sessions of individual CBT, each lasting 50 minutes. The CBT protocol includes standard therapeutic techniques such as ERP, cognitive restructuring, identification of maladaptive beliefs, psychoeducation, and relapse prevention strategies.

Control Group: Participants will be placed on a waiting list and will not receive any intervention during the active study period. CBT will be offered to these participants after study completion.

Participants in both groups will undergo comprehensive EEG assessments at three different time points: at baseline (pre-treatment), immediately following the CBT intervention (12 weeks post-baseline), and at a three-month follow-up (24 weeks post-baseline). EEG sessions will include:

Resting-State EEG (eyes closed):

Duration: 10-minute continuous recording.

Analysis Method: Low-Resolution Brain Electromagnetic Tomography (LORETA) to identify cortical activity patterns, specifically focusing on alpha-2 and beta frequency bands within regions implicated in OCD, such as the anterior cingulate cortex (ACC) and orbitofrontal cortex (OFC).

Emotional Oddball Paradigm:

Stimuli: Anxiety-provoking and neutral images or words presented randomly.

EEG measure: Event-Related Potentials (ERPs), particularly P300 amplitude and latency, to investigate attentional allocation and emotional processing alterations associated with OCD pathology and potential CBT-induced normalization.

Go/No-Go Task:

Purpose: Evaluate inhibitory control mechanisms and cognitive flexibility.

EEG measure: ERPs such as Error-Related Negativity (ERN), N2 (conflict monitoring), and P3 (response inhibition), known to be altered in OCD populations. This task will clarify whether CBT influences cognitive control functions at a neural level.

In addition to EEG, participants will complete several validated clinical measures at each time point to evaluate OCD symptom severity, anxiety, and depression levels. These scales include the Yale-Brown Obsessive-Compulsive Scale (Y-BOCS), Obsessive-Compulsive Inventory-Revised (OCI-R), Beck Depression Inventory-II (BDI-II), and Beck Anxiety Inventory (BAI).

EEG data will undergo rigorous preprocessing steps (bandpass filtering, independent component analysis for artifact removal, and segmentation into epochs) followed by ERP analysis using standardized software. Statistical comparisons will employ repeated measures ANOVA and linear mixed-effects models to identify significant differences between groups and across time points. Correlation analyses will examine the relationships between clinical improvements and neurophysiological changes observed via EEG.

Ultimately, this research aims to provide greater understanding of the biological processes underlying CBT effectiveness, potentially informing future targeted treatments and personalized therapeutic strategies for OCD.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 65 years
* Diagnosed with Obsessive-Compulsive Disorder (OCD) according to DSM-5 criteria
* Yale-Brown Obsessive Compulsive Scale (Y-BOCS) total score ≥16
* Not currently receiving psychiatric medication (at least 2-week washout required)
* No psychotherapy (including CBT) in the past 6 months
* Willing and able to participate in EEG procedures
* Capable of providing written informed consent

Exclusion Criteria:

* Use of any psychiatric medication in the past 2 weeks
* History of epilepsy, head trauma, or neurological disorders
* Current diagnosis of schizophrenia, bipolar disorder, or substance use disorder
* Severe physical illness or unstable medical condition
* Pregnancy or breastfeeding
* Prior CBT treatment for OCD within the past 6 months
* Currently participating in another clinical trial

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-10-25 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in OCD Symptom Severity on the Yale-Brown Obsessive Compulsive Scale (Y-BOCS) at Week 12 | Baseline, Week 12 (post-treatment), 3-month follow-up (Week 24)
  The Yale-Brown Obsessive Compulsive Scale (Y-BOCS) measures severity of obsessive-compulsive symptoms. The total score ranges from 0 (no symptoms) to 40 (extreme severity), with higher scores indicating greater OCD symptom severity.

SECONDARY OUTCOMES:
Change in ERP Component Amplitudes During EEG Tasks | Baseline, Week 12 (post-treatment), 3-month follow-up (Week 24)
  This outcome captures changes in Event-Related Potential (ERP) amplitudes recorded during cognitive tasks. Components include P300 amplitude during the emotional oddball task, and ERN, N2, and P3 amplitudes during the Go/No-Go task. These amplitudes are measured in microvolts (µV) and reflect neural responses to emotional and inhibitory stimuli.
Changes in Resting-State EEG Brain Activity | Baseline, Week 12 (post-treatment), 3-month follow-up (Week 24)
  Differences in resting-state EEG activity (LORETA-based cortical activity in alpha-2 and beta bands in ACC and OFC) from baseline to post-treatment and follow-up.
Change in Depression Symptoms | Baseline, Week 12 (post-treatment), 3-month follow-up (Week 24)
  Change from baseline in depressive symptoms as measured by Beck Depression Inventory-II (BDI-II). Scores range from 0 (minimal depression) to 63 (severe depression), with higher scores indicating greater depressive symptomatology.
Change in Anxiety Symptoms | Baseline, Week 12 (post-treatment), 3-month follow-up (Week 24)
  Change from baseline in anxiety levels measured by Beck Anxiety Inventory (BAI). Scores range from 0 (minimal anxiety) to 63 (severe anxiety), higher scores indicate greater anxiety severity.
Change in ERP Component Latencies During EEG Tasks | Baseline, Week 12 (post-treatment), 3-month follow-up (Week 24)
  This outcome captures changes in Event-Related Potential (ERP) latencies recorded during EEG-based cognitive tasks. Latencies of P300 (emotional oddball task), and N2 and P3 (Go/No-Go task) will be assessed. Measured in milliseconds (ms), these values reflect the timing of cognitive-emotional responses.

CONTACTS AND LOCATIONS:
Overall Officials: Eda Yılmazer, Phd, Principal Investigator — Beykoz University; Metin Çınaroğlu, Phd, Principal Investigator — Istanbul Nisantasi University
Locations (1):
- Üsküdar University, Istanbul, Turkey (Türkiye)